CLINICAL TRIAL: NCT05369793
Title: Clinical Study Evaluating the Safety and Efficacy of Roflumilast in Type 2 Diabetic Patients With Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Asmaa Elshafey Elsharab, Pharm D, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35420/4/22
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes (Adult Onset); Diabetic Neuropathies
Keywords: diabetes mellitus; diabetic neuropathy; hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Neuropathies; Diabetes Mellitus; Hyperglycemia | interventions — Thioctic Acid; Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha-lipoic acid arm (Active Comparator): Administration of alpha-lipoic acid 600 mg orally once daily for 3 months.
  Interventions: Drug: Alpha lipoic acid
- Roflumilast arm (Experimental): Administration of roflumilast 500 mcg orally once daily for 3 months.
  Interventions: Drug: Roflumilast

INTERVENTIONS:
Drug: Alpha lipoic acid — Administration of alpha-lipoic acid 600mg plus vildagliptin/metformin combination (50/1000mg) orally once daily for 3 months.
  Arms: Alpha-lipoic acid arm
Drug: Roflumilast — Administration of 500 mcg plus vildagliptin/metformin combination(50/1000mg) orally once daily for 3 months.
  Arms: Roflumilast arm

SUMMARY:
Evaluation of the side effects and efficacy of roflumilast on glycemic parameters, insulin resistance, oxidative and inflammatory markers in Type 2 diabetic patients with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of type 2 diabetes mellitus (T2DM).
* HbA1c at baseline: ≥7.5 % to 8.5 %.
* BMI between ≥26 and ≤35 kg/ m2.
* Established Diabetic neuropathy diagnosed by nerve conduction study (NCS).

Exclusion Criteria:

* Patients diagnosed with type 1 diabetes mellitus or diabetes secondary to pancreatitis or resection of the pancreas.
* Patients diagnosed with hemoglobinopathies, hemolytic anemia, or other diseases which interfere with HbA1c measurement.
* Thyroid disease, cardiovascular disease, peripheral vascular disease, coagulopathy, moderate to severe liver disease (bilirubin>1.5mg), or renal excretion ≤90ml/min.
* Patients on medications which can result in a change of weight (orlistat, metformin, clozapine, gabapentin) and patients on medications that can interfere with glucose or lipid metabolism (corticosteroids, non-selective β-blockers, thiazides, etc.)
* Treatment with any diabetes medications other than glimepiride prior to intervention.
* Clinically significant cardiac abnormalities (diagnosed clinically, history, or by X-ray/ECG) that were not related to type 2 diabetes mellitus and that required further evaluation.
* Patients with morbid obesity (BMI ≥ 40 kg/ m2).
* History or current diagnosis of major depressive disorders or other psychiatric disorders.
* Pregnant and breastfeeding women.
* Patients with any inflammatory diseases.
* Patients on cytochrome P450 inducers (e.g., rifampicin, phenobarbital, carbamazepine, phenytoin, etc.).
* Patients with Low vitamin B12 levels according to suggested normal values for T2DM patients over 60 years old (<400 pmol/L).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Change in fasting blood glucose | baseline and 3 months later
  Using glucose oxidase method for assessment of blood glucose and subtracting pre-treatment from post-treatment values
Change in plasma insulin level | baseline and 3 months later
  Subtracting pre-treatment from post-treatment values of plasma insulin
Change in HOMA-IR index | baseline and 3 months later
  HOMA-IR will be calculated for all patients at baseline and 3 months later.
Change in HOMA-B index | baseline and 3 months later.
  HOMA-B will be calculated for all patients at baseline and 3 months later.
Change in HbA1c | baseline and 3 months later
  Subtracting pre-treatment from post-treatment values of HbA1C

SECONDARY OUTCOMES:
Changes in TNF-alfa serum level | baseline and 3 months later
  Subtracting pre-treatment from post-treatment values of TNF-alfa.
Changes in malondialdehyde serum level (MDA) | baseline and 3 months later
  Subtracting pre-treatment from post-treatment values of MDA.
Changes in neurotensin serum levels | baseline and 3 months later
  Subtracting pre-treatment from post-treatment values of neurotensin serum levels.
Ewing score | baseline and 3 months later
  Subtracting pre-treatment from post-treatment changes in summation of the cardiac autonomic reflex tests (CARTs) including heart response to a deep breathing test, changes in immediate heart rate response to standing, and changes in blood pressure response to sustained handgrip testing.
Changes of Michigan Neuropathy Screening Instrument | baseline and 3 months later
  A 15-item questionnaire (MNSIQ) is used to assess deformation, infection, skin thickening of the skin's stratum corneum, and ulcers.
  MNSIQ was designed to screen for diabetic neuropathy through questionnaires on 15 questions that are related to neuropathic symptoms (pain, temperature, and sensation). Two of 15 (number 4 and 10) are vascular symptoms and are excluded from the total score regardless of the results. If you answered 'No' to questions 7 and 13, you will get 1 point. In the end, scores ranging from 0 to 13 indicate that the higher the score, the more severe the neuropathic symptoms.
Changes of Michigan Neuropathy Screening Instrument(MNSIE) | baseline and 3 months later
  A foot test (MNSIE) is used to assess deformation, infection, skin thickening of the skin's stratum corneum, and ulcers.
  MNSIE evaluates foot shape, foot ulceration, ankle reflex, sense of vibration of big toe, monofilament right and left. The score ranges from point 0 to 10, and when the score is above 2, it is diagnosed as neuropathy.
Changes of Douleur Neuropathique-4 (DN4) questionnaire (DN4) | baseline and 3 months later
  DN4 Neuropathic Pain Diagnostic Questionnaire which reflect positive symptoms for pain ( burning, painful cold, electric shocks, )

OTHER OUTCOMES:
Assessment of changes in patients' quality of life | baseline and 3 months later
  Using Diabetes Quality Of Life questionnaire (DQOL)
Major adverse cardiovascular events (MACE) | 3 months
  Major adverse cardiovascular events (MACE) as non-fatal myocardial infarction (MI), non-fatal stroke, and cardiovascular death.

CONTACTS AND LOCATIONS:
Locations (1):
- Asmaa Elshafey Elsharab, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elsharab A, Nooh MZ, Matard RS, Mostafa TM, El-Afify DR. Efficacy and Safety of Roflumilast versus Alpha-Lipoic Acid in Type 2 Diabetes with Neuropathy: A Comparative Clinical Study. Diabetes Metab Syndr Obes. 2025 Nov 13;18:4193-4210. doi: 10.2147/DMSO.S548285. eCollection 2025. PMID 41256904